CLINICAL TRIAL: NCT02206243
Title: An Observational Study to Evaluate the Safety and Efficacy of Embozene® Microspheres for Prostatic Arterial Embolization in Patients With Symptomatic Benign Prostatic Hyperplasia
Brief Title: Embozene® Microspheres for Prostatic Arterial Embolization in Patients With Symptomatic Benign Prostatic Hyperplasia
Acronym: EmboProstate
Status: Completed | Type: Observational
Sponsor: Jena University Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 3952-12/13
Record Dates: First submitted 2014-07-29; First posted 2014-08-01 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2017-11

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign prostatic hyperplasia; BPH
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Embozene: Patients receiving Embozene microspheres
  Interventions: Drug: Embozene Microspheres

INTERVENTIONS:
Drug: Embozene Microspheres — Intraarterial application
  Other Names: Vascular embolization

SUMMARY:
The purpose of this observational study is to evaluate the prostatic arterial embolization (PAE) with Embozene® Microspheres (Boston Scientific) in sphere sizes of 250 µm for the treatment of symptomatic benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
EmboProstate is an observational study that collects data of patients with benign prostatic hyperplasia that are treated with 250 µm Embozene ® Microspheres (Boston Scientific). The study evaluates the efficacy and safety of the microspheres for prostatic arterial embolization for benign prostata hyperplasia treatment. 10 adult male subjects will be enrolled in this study. If eligible patients are recruited, they will undergo the prostate artery embolization procedure in our radiology department. Once the catheter is placed in the prostate artery, a fluid containing thousands of tiny particles (microspheres) is injected through the catheter into these small arteries which nourish the prostate. The injected embospheres will slow the blood flow to the prostate reducing urinary tract symptoms caused by BPH. Within one week after PAE as well as after one, three and six months post-procedure an MRI examination ill occur. A follow-up visit using a questionnaire is due after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* male
* adults > 40 years old
* severe symptomatic BPH with IPSS > 18 and/or QoL > 3 or maximum urinary flow rate (Qmax) ≤ 15 ml/sec or transurethral catheter for retention
* no improvement after or intolerance of medical treatment for at least six months
* prostatic volume > 30 cm³

Exclusion Criteria:

* female
* less than 40 years old
* eGFR < 45 ml/min * m²
* suspicion of prostatic malignancy
* prostatic malignancy
* acute prostatitis or cystitis
* hydronephrosis
* bladder stone or bladder diverticulum
* urethral stenosis
* major surgery within 4 weeks prior to the screening visit
* active clinically serious infection
* progressive arteriosclerosis
* contraindications against angiography

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic (within clinical routine)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Symptomatic improvement of BPH symptoms (= International Prostate Symptom Score (IPSS) < 18 and reduction > 25% QoL (Quality of Life) < 4 & reduction ≥ & / or Qmax > 15 ml/s & increase of Qmax ≥ 3,0ml/s) at 6 and 12 months post intervention | Baseline, follow-up after 1 months, 6 months, 12 months, 24 months
  Improvement of feeling of incomplete bladder emptying, frequency, intermittency, urgency, weak stream, straining and nocturia

SECONDARY OUTCOMES:
Evaluate the safety of prostate artery embolization (PAE) for the treatment of lower urinary tract symptoms (LUTS) attributed to benign prostatic hyperplasia (BPH) | Within 1st week after PAE and follow-up after 1 months, 6 months, 12 months, 24 months
  The number and the severity of adverse events will be recorded to evaluate the safety of prostate artery embolization. Events will be reported by subjects within the 1st week after PAE and at follow-up after 6 months.

OTHER OUTCOMES:
Change in Qmax (reduction of postvoid residual volume) | Follow-up after 6 months
  Measure of urine flow rate. Q max = max flow rate
Reduction of prostate volume determined by volumetric measurement (MRI / transrectal Ultrasound) | Follow up MRI examinations: within the first week after PAE, 1, 3 and 6 months after PAE
  Measuring the percentage of prostate tissue devascularized, based on contrast-enhanced MRI by estimating the prostate volume and the estimated portion that is non-perfused on MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Teichgräber, Prof., Study Director — Institute of Diagnostic and Interventional Radiology; Marc-Oliver Grimm, Prof., Study Chair — Department of Urology; Tobias Franiel, Dr. med., Principal Investigator — Institute of Diagnostic and Interventional Radiology
Locations (1):
- Department of Radiology, University Hospital Jena, Jena, Thuringia, Germany